CLINICAL TRIAL: NCT00319020
Title: An Open Label, Long-term, Safety, and Tolerability Extension Study Using the Pediatric Formulation of Bosentan in the Treatment of Children With Idiopathic or Familial Pulmonary Arterial Hypertension Who Completed FUTURE 1
Brief Title: Bosentan in Children With Pulmonary Arterial Hypertension Extension Study
Acronym: FUTURE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-367; 2005-001967-70 (EudraCT Number)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: bosentan; pulmonary arterial hypertension; children; FUTURE 1
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bosentan (Experimental): Bosentan was administered at 4 mg/kg twice daily (b.i.d.) until the end of the study. It could be down-titrated to 2 mg/kg b.i.d. if not well tolerated.
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — 32-mg dispersible and breakable tablet. The body weight-adjusted dose of the dispersible tablet was dispersed in a teaspoon of water (not mixed with food) before being administered orally
  Other Names: Ro 47-0203; Tracleer

SUMMARY:
The main objective of the FUTURE 2 study was to assess the long-term safety and tolerability of the pediatric formulation of bosentan in children with idiopathic pulmonary arterial hypertension or familial pulmonary arterial hypertension who completed FUTURE 1 study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the parents or the legal representatives.
* Patients who completed the FUTURE 1 study.
* Patients who tolerated bosentan pediatric formulation and for whom bosentan is considered beneficial at the end of FUTURE 1.
* Males or females >= 2 and < 12 years of age at enrollment in FUTURE 2 (this study). Females who are menstruating must have a negative pregnancy test. A reliable method of contraception must be considered, if appropriate.

Exclusion Criteria:

* Intolerance to bosentan despite dose reductions.
* Any clinically significant laboratory abnormality that precludes continuation of bosentan therapy.
* Pregnancy or breast-feeding.
* Known hypersensitivity to bosentan or any of the excipients.
* Premature and permanent study drug discontinuation during FUTURE 1.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2005-08-23 (Actual); Primary Completion 2011-10-28 (Actual); Study Completion 2011-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andjela Kusic-Pajic, MD, Study Director — Actelion

REFERENCES:
- [Result] Berger RM, Haworth SG, Bonnet D, Dulac Y, Fraisse A, Galie N, Ivy DD, Jais X, Miera O, Rosenzweig EB, Efficace M, Kusic-Pajic A, Beghetti M. FUTURE-2: Results from an open-label, long-term safety and tolerability extension study using the pediatric FormUlation of bosenTan in pUlmonary arterial hypeRtEnsion. Int J Cardiol. 2016 Jan 1;202:52-8. doi: 10.1016/j.ijcard.2015.08.080. Epub 2015 Aug 9. PMID 26386921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 Children ( >= 2 years and < 12 years) with idiopathic or familial pulmonary arterial hypertension were recruited from 11 centers across Europe and USA and enrolled in the FUTURE 1 trial (baseline). Only patients who completed FUTURE 1 (n=34) could be enrolled in FUTURE 2. Enrollment in FUTURE 2 started August 23, 2005.
Pre-assignment Details: The actual number of patients enrolled in FUTURE 2 (F-2) was 33 because 2 patients did not complete FUTURE 1 (F-1) and one patient completed F-1 but was not enrolled in F-2.
Groups:
- Patients With Previous Bosentan: This group included patients who already received bosentan (film-coated tablets) before enrollment in FUTURE 1, and then received the pediatric formulation of bosentan (dispersible tablets) during FUTURE 1 and FUTURE 2 (initiatied at 2 mg/kg b.i.d. for 4 weeks, then up-titrated to the maintenance dose of 4 mg/kg b.i.d. for the next 8 weeks of the FUTURE 1 trial (AC-052- 365) and to be continued in FUTURE 2. The dose could be down-titrated to 2 mg/kg b.i.d. if not tolerated).
  Note: In this single arm trial, data are presented according to whether patients received bosentan or not before enrollment in FUTURE 1 but all the subjects received the study drug according to the same regimen.
- Bosentan-naive Patients: This group included patients who were not treated with bosentan before enrollment in FUTURE 1, and received the pediatric formulation of bosentan (dispersible tablets) during FUTURE 1 and FUTURE 2 according to the same dosing regimen as described for "Patients with previous bosentan".
  Note: In this single arm trial, data are presented according to whether patients received bosentan or not before enrollment in FUTURE 1 but all the subjects received the study drug according to the same regimen.
Period: Overall Study
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients
Started | 15 | 21
Enrollment in FUTURE 2 (F-2) | 13 | 20
Completed | 8 | 8
Not Completed | 7 | 13
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — F-1 completed but not enrolled in F-2 | 1 | 0
Not completed — Administrative reason | 0 | 5
Not completed — Disease progression | 0 | 2
Not completed — Transplant | 0 | 1
Not completed — Treatment failure | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With Previous Bosentan: This group included patients who already received bosentan (film-coated tablets) before enrollment in FUTURE 1, and then received the pediatric formulation of bosentan (dispersible tablets) during FUTURE 1 and FUTURE 2 (initiation at 2 mg/kg b.i.d. for 4 weeks, then up-titrated to the maintenance dose of 4 mg/kg b.i.d. for the next 8 weeks of the FUTURE 1 trial (AC-052- 365) and to be continued in FUTURE 2. The dose could be down-titrated to 2 mg/kg b.i.d. if not tolerated).
- Total: Total of all reporting groups
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Continuous [Median (Full Range); unit: Years] | 7 [3 to 10] | 7 [2 to 11] | 7 [2 to 11]
Age, Customized [Number; unit: Participants]
  2-3 years old | 1 | 3 | 4
  4-5 years old | 3 | 6 | 9
  6-11 years old | 11 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 10 | 11 | 21
Etiology of pulmonary arterial hypertension (PAH) [Number; unit: Participants] — Children included in the study had a diagnosis of pulmonary arterial hypertension (PAH) belonging to one of the following two categories: 1- Idiopathic PAH, 2- Familal PAH
  Participants
    Idiopathic PAH | 12 | 19 | 31
    Familial PAH | 3 | 2 | 5
Duration of pulmonary arterial hypertension (PAH) [Median (Full Range); unit: Months] | 37.6 [1.2 to 82.6] | 14 [0 to 133.5] | 25.8 [0 to 133.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study (EOS) in Height for Age.
Description: In order to compare the growth data with those of healthy children, growth curves are calculated from height data collected throughout the follow-up period. For each patient, height measured at each study visit was converted to a z-score and expressed in standard deviations (SD) from WHO growth standards. The Z-score was calculated according to the following formula:
  Z-score = (observed value of the study participant - median value of the reference population) / SD value of the reference population
Time Frame: From baseline (FUTURE 1) up to 28 days after study treatment discontinuation (EOS or premature study treatment discontinuation), i.e. 32 months in average
Population: All-treated analysis set (all patients who received at least one dose of study drug in the combined FUTURE 1 / FUTURE 2 trial periods). Missing or incomplete data were treated as missing.
Measure: Median (Full Range); unit: Z-score
Groups:
- Patients With Previous Bosentan: This group included patients who already received bosentan (film-coated tablets) before enrollment in FUTURE 1, and then received the pediatric formulation of bosentan (dispersible tablet) during FUTURE 1 and FUTURE 2 (initiation at 2 mg/kg b.i.d. for 4 weeks, then up-titrated to the maintenance dose of 4 mg/kg b.i.d. for the next 8 weeks of the FUTURE 1 trial (AC-052- 365) and to be continued in FUTURE 2. The dose could be down-titrated to 2 mg/kg b.i.d. if not tolerated).
- Bosentan-naive Patients: This group included patients who were not treated with bosentan before enrollment in FUTURE 1, and received the pediatric formulation of bosentan (dispersible tablet) during FUTURE 1 and FUTURE 2 according to the same dosing regimen as described for "Patients with previous bosentan".
  Note: In this single arm trial, data are presented according to whether patients received bosentan or not before enrollment in FUTURE 1 but all the subjects received the study drug according to the same regimen.
- Total: All patients (bosentan-naive patients and patients treated with film-coated bosentan tablets before enrollment) who received at least one dose of study drug (bosentan dispersible tablets) in the combined FUTURE 1 / FUTURE 2 trial periods.
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 10 | 14 | 24
Z-score
  Z-score at baseline | -0.8 [-3.32 to 3.72] | 0.32 [-2.62 to 1.99] | -0.64 [-3.32 to 3.72]
  Z-score at EOS | -0.74 [-3.52 to 2.78] | -0.08 [-2.44 to 1.84] | -0.36 [-3.52 to 2.78]
  Z-score change from baseline to EOS | -0.05 [-0.94 to 0.91] | -0.01 [-0.77 to 1.08] | -0.01 [-0.94 to 1.08]

2. Primary Outcome: Change From Baseline to End of Study (EOS) in Body Weight
Description: The main study objective was to assess the long-term safety and tolerability of bosentan in children with PAH, including growth as measured by changes from baseline in body weight and height.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: kg
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 10 | 14 | 24
kg
  Weight at baseline | 19.6 [12.5 to 30.2] | 21.6 [11 to 39] | 19.6 [11 to 39]
  Weight change from baseline to EOS | 8.2 [5 to 24.8] | 8.5 [1.8 to 18.5] | 8.3 [1.8 to 24.8]

3. Primary Outcome: Change From Baseline to End of Study (EOS) in Systolic Blood Pressure (SBP)
Description: The main study objective was to assess the long-term safety and tolerability of bosentan in children with PAH, including changes from baseline in blood pressure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 10 | 14 | 24
mmHg
  SBP at baseline | 101.5 [87 to 115] | 104 [79 to 121] | 102.5 [79 to 121]
  SBP change from baseline to EOS | -10.5 [-20 to 25] | 4 [-21 to 28] | -4.5 [-21 to 28]

4. Primary Outcome: Change From Baseline to End of Study (EOS) in Diastolic Blood Pressure (DBP)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 10 | 13 | 23
mmHg
  DBP at baseline | 54.5 [47 to 94] | 60 [52 to 75] | 59 [47 to 94]
  DBP change from baseline to EOS | -5 [-34 to 19] | -2 [-13 to 20] | -3 [-34 to 20]

5. Primary Outcome: Change From Baseline to End of Study (EOS) in Pulse Rate
Description: The main study objective was to assess the long-term safety and tolerability of bosentan in children with PAH, including changes from baseline in pulse rate.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Beats per minutes
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 11 | 14 | 25
Beats per minutes
  Pulse rate at baseline | 87 [55 to 118] | 94.5 [62 to 133] | 88 [55 to 133]
  Pulse rate change from baseline to EOS | -11 [-46 to 36] | -10 [-30 to 11] | -11 [-46 to 36]

6. Primary Outcome: Proportion of Patients With Treatment-emergent Liver Function Abnormalities
Description: The main study objective was to assess the long-term safety and tolerability of bosentan in children with PAH, including laboratory abnormalities related to liver enzymes.
  Proportion of patients with increase in alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above 3 times upper limit of normal (ULN) is reported here.
Time Frame: After baseline, up to 1 calendar day after study treatment discontinuation in FUTURE 1 or FUTURE 2, i.e. 31 months in average
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 15 | 21 | 36
Percentage of participants
  ALT > 3 x ULN | 0 | 4.8 | 2.8
  AST > 3 x ULN | 0 | 4.8 | 2.8

7. Primary Outcome: Proportion of Patients With Treatment-emergent Hemoglobin Abnormalities
Description: The main study objective was to assess the long-term safety and tolerability of bosentan in children with PAH, including hemoglobin abnormalities.
  Proportion of patients with marked hemoglobin decreases (i.e., decrease of or above 15% of the lower normal limit (LL)) is reported here.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 15 | 21 | 36
Percentage of participants | 13.3 | 9.5 | 11.1

8. Primary Outcome: Number of Subjects With Adverse Events Leading to Premature Discontinuation of Study Treatment
Time Frame: From the first study drug administration in FUTURE 1, for an average of 31 months
Measure: Number; unit: Participants
Arm/Group | Patients With Previous Bosentan | Bosentan-naive Patients | Total
Number analyzed (Participants) | 15 | 21 | 36
Participants | 1 | 5 | 6

ADVERSE EVENTS:
Time Frame: From the first administration of study treatment and for an average of 31 months for frequent adverse events (up to 1 day after study treatment discontinuation), and for an average of 32 months (up to 28 days after study treatment discontinuation) for serious adverse events
Groups:
- Patients With Previous Bosentan: Patients who already received bosentan (film-coated tablets) before enrollment in FUTURE 1, and then received the pediatric formulation of bosentan during FUTURE 1 / FUTURE 2
- Bosentan_naive Patients: Patients who were not treated with bosentan before enrollment in FUTURE 1, and received the pediatric formulation of bosentan during FUTURE 1 / FUTURE 2
- Single Arm Bosentan_Total: All patients included in Future 1 / FUTURE 2 whether they received bosentan or not bosentan before enrollment in FUTURE 1
Arm/Group | Patients With Previous Bosentan | Bosentan_naive Patients | Single Arm Bosentan_Total
Serious Adverse Events (participants affected / at risk) | 9/15 | 9/21 | 18/36
Other Adverse Events (participants affected / at risk) | 12/15 | 16/21 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Previous Bosentan (N=15) | Bosentan_naive Patients (N=21) | Single Arm Bosentan_Total (N=36)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ADENOIDECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
ARTERIAL CATHETERISATION (Investigations) | 0 (0) | 1 (1) | 1 (1)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BALLOON ATRIAL SEPTOSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
CATHETERISATION CARDIAC (Investigations) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 2 (6) | 3 (7)
DIAPHRAGMATIC HERNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
DYSTONIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
INJECTION SITE NODULE (General disorders) | 0 (0) | 1 (1) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
MEDICAL DEVICE COMPLICATION (General disorders) | 0 (0) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (4)
PULMONARY ARTERIAL PRESSURE (Investigations) | 0 (0) | 1 (1) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
PULMONARY VEIN STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
SYSTEMIC-PULMONARY ARTERY SHUNT (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Previous Bosentan (N=15) | Bosentan_naive Patients (N=21) | Single Arm Bosentan_Total (N=36)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 5 (6) | 6 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (4)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 1 (2) | 2 (3)
AGGRESSION (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 1 (1) | 2 (3) | 3 (4)
BRONCHITIS (Infections and infestations) | 2 (2) | 3 (4) | 5 (6)
CHEST PAIN (General disorders) | 0 (0) | 3 (10) | 3 (10)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 2 (4)
CYANOSIS (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (3) | 3 (4)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 2 (3)
ENURESIS (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
FATIGUE (General disorders) | 0 (0) | 2 (3) | 2 (3)
FLUSHING (Vascular disorders) | 1 (1) | 3 (4) | 4 (5)
H1N1 INFLUENZA (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 3 (6) | 4 (7)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 3 (4)
NASOPHARYNGITIS (Infections and infestations) | 3 (5) | 4 (6) | 7 (11)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
PALPITATIONS (Cardiac disorders) | 0 (0) | 2 (4) | 2 (4)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
PNEUMONIA (Infections and infestations) | 1 (5) | 2 (2) | 3 (7)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (4)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
PYREXIA (General disorders) | 1 (1) | 2 (2) | 3 (3)
SYNCOPE (Nervous system disorders) | 2 (2) | 1 (4) | 3 (6)
TONSILLITIS (Infections and infestations) | 1 (2) | 1 (1) | 2 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (6) | 5 (7)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
VOMITING (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
ALLERGY TO PLANTS (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
CATHETER SITE PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
NIPPLE SWELLING (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
PERTUSSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
TOOTH DISCOLOURATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related article or abstract written independently by investigators should be submitted to Actelion for review at least 60 days prior to submission for publication or presentation.